CLINICAL TRIAL: NCT03880461
Title: Cluster Randomized Trial of a Mobile Health Intervention to Achieve Appropriate Gestational Weight Gain in Overweight/Obese Women
Brief Title: A Mobile Health Intervention to Achieve Appropriate Gestational Weight Gain in Overweight/Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1352535-1
Record Dates: First submitted 2019-03-13; First posted 2019-03-19 (Actual); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-03

CONDITIONS: Gestational Weight Gain
Keywords: Gestational weight gain; Lifestyle; Intervention; Body weight; Overweight; Obesity; Signs and Symptoms; Body weight changes
MeSH Terms: conditions — Gestational Weight Gain; Body Weight; Overweight; Obesity; Signs and Symptoms; Body Weight Changes

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle Intervention (Experimental): The goal of the intervention is to help women achieve GWG within the range recommended by the Institute of Medicine. The lifestyle intervention will be delivered through 1 telephone counseling session with a study dietician trained in motivational interviewing techniques, as well as through technology-based tools, automated text messages and weekly e-mails of core lifestyle intervention sessions. Personalized text messages and 1:1 telephone coaching sessions will be given to those who are not meeting the GWG guidelines.
  Interventions: Behavioral: Lifestyle Intervention
- Usual Care - Control (No Intervention): Usual Medical Care

INTERVENTIONS:
Behavioral: Lifestyle Intervention — Behavioral lifestyle intervention
  Arms: Lifestyle Intervention

SUMMARY:
The aim of this trial is to investigate the effectiveness of a mobile health (mhealth) intervention to help overweight and obese women achieve appropriate gestational weight gain (GWG) for their pre-pregnancy body mass index (BMI). The goal of the intervention is to help women achieve GWG within the range recommended by the Institute of Medicine. The investigators propose an adaptive intervention that begins with an effective, yet low resource-intensive treatment and then provides incremental support and resources only to patients who need them. The intervention includes: 1) an mHealth tool allowing data to be automatically transmitted to a mobile website; 2) personalized text messages; and 3) personalized 1:1 telephone coaching sessions. The latter more intensive components are reserved for patients whose GWG is not within the IOM guidelines. The lifestyle intervention will be delivered through 1 telephone counseling session with a study dietician trained in motivational interviewing techniques, as well as through technology-based tools, automated text messages and weekly e-mails of core lifestyle intervention sessions. Personalized text messages and 1:1 telephone coaching sessions will be given to those who are not meeting the GWG guidelines. The lifestyle intervention will be compared to usual medical care. Maternal outcomes will be assessed shortly before delivery and at 6 weeks postpartum. Infant birthweight and weight at one year will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Women receiving prenatal care at Kaiser Permanente San Francisco and Oakland and whose obstetric care clinicians consent to participate;
* Pregravid BMI 25 to <40 (as determined from a measured pregravid weight in electronic medical record);
* Has access to a smartphone and Wi-Fi;
* Provides informed consent to participate.

Exclusion Criteria:

* Multiple births;
* Planning to move out of the area during the study period;
* Inability to speak, read, or understand English;
* Placed on bed rest at time of enrollment; ->15 weeks' gestation at enrollment.

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study is only enrolling female participants.
Enrollment: 1335 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Kaiser Permanente Oakland, Oakland, California
  - Kaiser Permanente Redwood City, Redwood City, California
  - Kaiser Permanente San Francisco, San Francisco, California
  - Kaiser Permanente Santa Clara, Santa Clara, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sridhar SB, Ferrara A, Brown SD, Quesenberry CP, Xu F, Liu E, Sedgwick T, Kissel P, Serrato Bandera HD, Albright C, Hedderson MM. Protocol of an adaptive mobile health intervention for the management of gestational weight gain: The LEAP cluster randomized controlled trial. Contemp Clin Trials. 2025 Feb;149:107781. doi: 10.1016/j.cct.2024.107781. Epub 2024 Dec 20. PMID 39710337

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Arm - PATIENTS: In addition to usual medical care, patients in the intervention arm will receive access to mHealth tools to manage gestational weight gain (GWG), including a scale, physical activity tracker, and smartphone application, and for those not meeting GWG guidelines, personalized text messages and personalized 1-1 coaching sessions.
- Usual Care Arm - PATIENTS: Patients in the usual care arm will receive the standard obstetric care offered at Kaiser Permanente Northern California.
Period: Overall Study
Arm/Group | Intervention Arm - PATIENTS | Usual Care Arm - PATIENTS
Started | 714 | 621
Completed | 645 | 560
Not Completed | 69 | 61
Not completed — Determined ineligible after enrollment | 45 | 44
Not completed — No weight measurement after enrollment | 24 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm - PATIENTS | Usual Care Arm - PATIENTS | Total
Number analyzed (Participants) | 714 | 621 | 1335
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (4.7) | 33.4 (4.5) | 33.4 (4.6)
Age, Customized [Count of Participants; unit: Participants]
  Age (years): 21 - 29 | 158 | 122 | 280
  Age (years): 30 - 34 | 259 | 238 | 497
  Age (years): 35 - 39 | 234 | 215 | 449
  Age (years): 40 - 46 | 63 | 46 | 109
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 714 | 621 | 1335
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race / Ethnicity: Non-Hispanic White | 237 | 211 | 448
  Race / Ethnicity: Black | 41 | 40 | 81
  Race / Ethnicity: Asian / Pacific Islander | 175 | 137 | 312
  Race / Ethnicity: Hispanic | 186 | 165 | 351
  Race / Ethnicity: Native American | 10 | 4 | 14
  Race / Ethnicity: Islander | 6 | 4 | 10
  Race / Ethnicity: Multiracial | 37 | 41 | 78
  Race / Ethnicity: Unknown / Missing | 22 | 19 | 41
Region of Enrollment [Number; unit: participants]
  United States | 714 | 621 | 1335
Pre-pregnancy BMI (Continuous) [Mean (Standard Deviation); unit: kg/m2] | 29.7 (3.8) | 30.0 (3.9) | 29.8 (3.8)
Pre-pregnancy BMI (Customized) [Count of Participants; unit: Participants]
  Overweight (25.0 - 29.9) | 430 | 354 | 784
  Obese (30.0 - 39.9) | 284 | 267 | 551
Parity (Customized) [Count of Participants; unit: Participants]
  Nulliparous | 319 | 238 | 557
  Primiparous | 270 | 239 | 509
  Multiparous | 103 | 127 | 230
  Unknown / Missing | 22 | 17 | 39

OUTCOME MEASURES:

1. Primary Outcome: Total Gestational Weight Gain (GWG)
Description: Calculated as last measured pregnancy weight at the time of delivery minus measured weight at 10 gestational weeks
Time Frame: From 10 gestational weeks until time of delivery (duration of up to 9 months)
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Intervention Arm - PATIENTS | Usual Care Arm - PATIENTS
Number analyzed (Participants) | 591 | 520
kilograms | 10.5 (5.7) | 11.3 (5.9)
Statistical Analysis 1: Comparison: Intervention Arm - PATIENTS vs Usual Care Arm - PATIENTS; Test type: Superiority; p = 0.014, t-test, 2 sided

2. Primary Outcome: Rate of Total GWG
Description: Calculated as total gestational weight gain / (# of weeks between 10 gestational weeks and the time of delivery)
Time Frame: From 10 gestational weeks until time of delivery (duration of up to 9 months)
Measure: Mean (Standard Deviation); unit: kilograms/week
Arm/Group | Intervention Arm - PATIENTS | Usual Care Arm - PATIENTS
Number analyzed (Participants) | 645 | 560
kilograms/week | 0.26 (0.17) | 0.28 (0.16)
Statistical Analysis 1: Comparison: Intervention Arm - PATIENTS vs Usual Care Arm - PATIENTS; Test type: Superiority; p = 0.003, t-test, 2 sided

3. Primary Outcome: Proportion of Women Meeting the Institute of Medicine's GWG Recommendation
Description: Proportion of women meeting the IOM's GWG recommendation for weekly rate of GWG
Time Frame: From 10 gestational weeks until time of delivery (duration of up to 9 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm - PATIENTS | Usual Care Arm - PATIENTS
Number analyzed (Participants) | 645 | 560
Participants | 172 | 126
Statistical Analysis 1: Comparison: Intervention Arm - PATIENTS vs Usual Care Arm - PATIENTS; Test type: Superiority; p = 0.108, ANOVA

4. Secondary Outcome: Trimester-specific Weekly Rate of GWG
Time Frame: 0 - 13 gestational weeks; 14 - 26 gestational weeks; 27 - 40 gestational weeks
Reporting Status: Not Posted

5. Secondary Outcome: GWG Trajectory Throughout Pregnancy
Time Frame: From 10 gestational weeks until time of delivery (duration of up to 9 months)
Reporting Status: Not Posted

6. Secondary Outcome: Change in Moderate to Vigorous Physical Activity (in MET Hrs/Week) as Assessed by the Pregnancy Physical Activity Questionnaire (PPAQ)
Description: We will assess change in moderate to vigorous physical activity between study assessments in pregnancy. The sports and exercise domain encompasses 10 PPAQ activities of moderate intensity (ranging 3.2 MET to 6 MET) and 2 PPAQ activities of vigorous intensity (6.5 MET and 7 MET). The volumes of all activities in the sports and exercise domain will be summed to arrive at an estimate of overall volume of moderate to vigorous intensity sports and exercise activity, expressed in MET hours per week. Higher levels of activity are generally associated with better outcomes. The distributions of all physical activity variables will be assessed for outliers.
Time Frame: Between 12 weeks and 33 weeks of pregnancy
Reporting Status: Not Posted

7. Secondary Outcome: Overall Diet Quality According to the Healthy Eating Index-2015 (HEI-2015)
Description: The HEI-2015 reflects adherence to the 2015-2020 Dietary Guidelines for Americans; it is comprised of 13 components as well as an overall score. The scoring system ranges from 0 to 100, where higher values indicate a better diet quality.
Time Frame: Assessed at 12 weeks of pregnancy
Reporting Status: Not Posted

8. Secondary Outcome: Postpartum Weight Retention
Time Frame: Assessed at 6 weeks postpartum
Reporting Status: Not Posted

9. Secondary Outcome: The Proportion of Infants With Appropriate Birthweight (>10th and <90th Percentile of Sex-, Gestational Age-, and Racial/Ethnic-specific Distribution)
Time Frame: Assessed at birth
Reporting Status: Not Posted

10. Secondary Outcome: Infant Growth (BMI Z-score)
Time Frame: From birth to 12 months of age
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse outcome data were collected during pregnancy from enrollment to delivery (duration of up to 9 months).
Arm/Group | Intervention Arm - PATIENTS | Usual Care Arm - PATIENTS
All-Cause Mortality (participants affected / at risk) | 0/714 | 0/621
Serious Adverse Events (participants affected / at risk) | 0/714 | 0/621
Other Adverse Events (participants affected / at risk) | 44/714 | 29/621
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Arm - PATIENTS (N=714) | Usual Care Arm - PATIENTS (N=621)
Total pregnancy loss or stillbirth (Pregnancy, puerperium and perinatal conditions) | 44 | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-26): https://cdn.clinicaltrials.gov/large-docs/61/NCT03880461/Prot_SAP_000.pdf